CLINICAL TRIAL: NCT03469726
Title: Diagnostic Accuracy of Contrast-enhanced Diffusion-weighted MRI for Liver Metastases of Pancreatic Cancer: Towards Adequate Staging and Follow-up of Pancreatic Cancer
Brief Title: Contrast-enhanced Diffusion-weighted MRI to Detect Liver Metastases in Patients With Pancreatic Cancer
Acronym: DIA-PANC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL60473.091.17
Record Dates: First submitted 2018-02-28; First posted 2018-03-19 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2020-10

CONDITIONS: Pancreatic Neoplasms
Keywords: Liver metastases; Diffusion weighted MRI
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: International multicenter prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with (suspected) PDAC (Other): Patients with (suspected) pancreatic cancer will undergo additional Contrast-enhanced Diffusion-weighted MRI (CE-DW-MRI) within two weeks from the CECT.
  Suspected liver lesions on CECT and/or CE-DW-MRI will be biopsied to obtain histopathology as reference standard. For liver lesions without histopathologic proof of metastases a paired follow-up CECT and CE-DW-MRI serve as a composite reference standard. Follow up CECT and CE-DW-MRI will be performed in all patients at 3, 6, and 12 months.
  Interventions: Diagnostic Test: Contrast-enhanced Diffusion-weighted MRI

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced Diffusion-weighted MRI — An MRI scan enhanced with intravenous contrast and with diffusion imaging at several B-values

SUMMARY:
Given the dismal prognosis of pancreatic cancer, detecting liver metastases early can avoid inappropriate therapy with the associated substantial risks, long-term hospital admissions and high costs, but without survival benefit. The current standard of diagnostic workup with contrast-enhanced CT (CECT) has a poor sensitivity (38-76%) for the detection of liver metastases. As more sophisticated and expensive treatment options emerge, better staging of pancreatic cancer is needed to avoid unnecessary procedures and select the most appropriate treatment strategy. New imaging modalities are available, but their value in staging of pancreatic cancer has not been evaluated yet. Therefore prospective imaging studies are necessary.

The main aim of this study is to determine the diagnostic accuracy of contrast-enhanced diffusion-weighted MRI (CE-DW-MRI) in the detection of liver metastases in patients with pancreatic cancer compared to a reference standard of histopathology and follow up imaging.

The study is an international, multicenter prospective cohort study (inclusion of patients until 138 patients with liver metastases are included, with a total maximum of 465 patients). Patients with pancreatic cancer will undergo additional CE-DW-MRI within two weeks from the CECT. CECT and CE-DW-MRI will be read independently by two radiologists. Suspected liver lesions on CECT and/or CE-DW-MRI will be biopsied to obtain histopathology as reference standard. For liver lesions without histopathologic proof of metastases a paired follow-up CECT and CE-DW-MRI serve as a composite reference standard. Pancreatic resection will be pursued in patients without proven liver or distant metastases. Patients with locally advanced or metastatic disease will be offered palliative treatment. Follow up CECT and CE-DW-MRI will be performed in all patients at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* clinical suspicion of pancreatic cancer
* written (signed and dated) informed consent

Exclusion Criteria:

* previous treatment for pancreatic cancer (e.g. chemotherapy, radiotherapy, surgery, ablation therapy)
* concomitant malignancies, except for adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri. Subjects with prior malignancies must be disease-free for at least 5 years
* contra-indications to undergo CT (due to e.g. extreme claustrophobia, untreatable contrast allergy, renal function impairment)
* contra-indications to undergo MRI (due to e.g. claustrophobia, untreatable contrast allergy, or not MRI compatible medical devices)
* insufficient command of the Dutch language to be able to understand the patient information or fill in the questionnaires
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Estimated)
Dates: Start 2017-12-22 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of CE-DW-MRI | Baseline
  Sensitivity and Specificity of CE-DW-MRI for the detection of liver metastases in patients with pancreatic cancer compared to CECT.

SECONDARY OUTCOMES:
Detection of metastasis on CE-DW-MRI in follow-up (3, 6 and 12 months after baseline) | 3, 6 and 12 months
  Detection of metastasis with CE-DW-MRI, compared to CECT, in follow-up (3, 6 and 12 months after baseline) of patients with pancreatic cancer, after or during therapy
Assess local resectability | Baseline
  Sensitivity and specificity for CT and MRI to assess local resectability for all patients that underwent surgery

OTHER OUTCOMES:
One year survival | Maximum 1 year
  Survival rate after 1 year of follow-up
Median survival | Maximum 1 year
  Median survival time
Disease free survival | Maximum 1 year
  Time without (local) recurrence of cancer in patients that underwent resection
Progression free survival | Maximum 1 year
  Time without progression of cancer

CONTACTS AND LOCATIONS:
Overall Officials: John J. Hermans, dr. ir., Principal Investigator — Radboudumc, Department of Radiology and Nuclear Medicine; Kees C.J.H.M. van Laarhoven, prof. dr., Principal Investigator — Radboudumc, Department of Surgery
Locations (7):
- Konstantopouleio general hospital, Athens, Greece
- Netherlands (4):
  - Radboudumc, Nijmegen, Gelderland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Medisch Spectrum Twente, Enschede
  - Universitair Medisch Centrum Groningen, Groningen
- Hospital Universitario Ramón y Cajal, Madrid, Spain
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Litjens G, Riviere DM, van Geenen EJM, Radema SA, Brosens LAA, Prokop M, van Laarhoven CJHM, Hermans JJ. Diagnostic accuracy of contrast-enhanced diffusion-weighted MRI for liver metastases of pancreatic cancer: towards adequate staging and follow-up of pancreatic cancer - DIA-PANC study: study protocol for an international, multicenter, diagnostic trial. BMC Cancer. 2020 Aug 10;20(1):744. doi: 10.1186/s12885-020-07226-0. PMID 32778061